CLINICAL TRIAL: NCT03362216
Title: Clinical Efficacy and Safety of Compound Methyl Salicylate Liniment in the Treatment of Acute and Chronic Soft Tissue Pain：a Multicenter, Randomized, Positive Controlled Clinical Trial
Brief Title: Clinical Efficacy and Safety of Compound Methyl Salicylate Liniment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, baoguojiang, Dean of Peking University People's Hospital, Director of department of orthopaedic surgery of Peking University, Chairman of China trauma rescue&treatment association, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUPH20170999
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Soft Tissue Injuries
Keywords: soft tissue, pain
MeSH Terms: conditions — Soft Tissue Injuries; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Treated with Compound Methyl Salicylate Liniment group
  Interventions: Drug: Compound Methyl Salicylate Liniment
- Control group (Active Comparator): Treated with Diclofenac Sodium Liniment group
  Interventions: Drug: Diclofenac Sodium Liniment

INTERVENTIONS:
Drug: Compound Methyl Salicylate Liniment — Compound Methyl Salicylate Liniment, apply to the affected area, 3 times a day.Course of treatment: 7 days
  Arms: experimental group
Drug: Diclofenac Sodium Liniment — Diclofenac Sodium Liniment, apply to the affected area, 3 times a day. Course of treatment: 7 days
  Arms: Control group

SUMMARY:
This clinical trial program was established according to the ethical principles of the Helsinki declaration and the GCP guiding principle, and a randomized grouping method was used to evaluate the efficacy and safety of Compound Methyl Salicylate Liniment in the treatment of acute and chronic soft tissue pain with a positive control drug, named Diclofenac Sodium Liniment.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, parallel controlled multicenter clinical trial for evaluate the efficacy and safety of Compound Methyl Salicylate Liniment in the treatment of acute and chronic soft tissue pain with a positive control drug, named Diclofenac Sodium Liniment. A total of 216 participants with acute or chronic tissue pain participated in this clinical trial. The clinical trial cases were equally allocated to each research center, and each center had 30-35 cases. The proportion of patients with acute soft tissue pain and chronic soft tissue pain was 1:1, and the proportion of the experimental group and the control group was 1:1.The observation index include self pain scale record, tenderness scale and swelling, the evaluation period was 7 days.

The statistical analysis plan is prepared by the unit responsible for the statistics, and is prepared before the formal analysis of the data, and is discussed and identified at the blind audit meeting with the major researchers. Statistical analysis will use SAS8.2 statistical analysis software for data processing, and other statistical analysis plan to make detailed provisions. All the statistical tests were two-sided, and the value of P was less than or equal to 0.05, which would be considered statistically significant. Measurement data use case number, mean, standard deviation, minimum, maximum, median and four sub spacing description, counting data and grade data use case number, percentage description.

ELIGIBILITY:
Inclusion Criteria:

* Patients with various causes of acute and chronic soft tissue
* Local symptoms and signs include pain, swelling, bruising, tenderness, joint dysfunction; X-ray showed no fracture, dislocation, bone tumors and bone metabolism and open injury.

Exclusion Criteria:

* Patients who do not belong to the scope of drug use
* Muscle, tendon, ligament and other soft tissue have broken completely
* Accompanied by skin damage or fracture, joint dislocation, bone tumor and metabolic bone disease local tissue damage
* Use of other drugs or therapies for the treatment of acute and chronic soft tissue pain after trauma
* Difficult to evaluate the effectiveness and safety of new drugs
* Severe hypertension, severe heart and lung dysfunction, severe arrhythmia, liver, kidney, hematopoietic system and other serious primary diseases, mental patients
* Pregnant women, lactating women
* Allergic constitution and allergic to the known components of the drug
* Participated in other clinical trials in the past month
* Use similar analgesics within a week
* Other researchers considered inappropriate patients to participate in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-04-07 (Actual); Primary Completion 2009-05-22 (Actual); Study Completion 2009-06-12 (Actual)

PRIMARY OUTCOMES:
Main observation index | 7 days
  Self pain scale record (VAS). A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.

SECONDARY OUTCOMES:
Secondary observation index | 7 days
  Record of tenderness scale(VAS), Swelling. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.

CONTACTS AND LOCATIONS:
Overall Officials: People's Hospital Peking University, Study Director — Peking University

IPD SHARING:
Plan to Share IPD: No